CLINICAL TRIAL: NCT04526639
Title: Virtual Reality-based Rehabilitation for Pediatric TBI (R00 Phase)
Brief Title: VR Cognitive Rehabiliation for Pediatric TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Lowell (Other)
Collaborators: Spaulding Rehabilitation Hospital (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Jiabin Shen, PhD, Assistant Professor, Psychology, University of Massachusetts, Lowell
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R00HD093814 (NIH)
Record Dates: First submitted 2020-08-18; First posted 2020-08-26 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality games for training executive functions (Experimental): Virtual Reality games for training three core executive functions
  Interventions: Behavioral: Virtual Reality-based Interactive Cognitive Training Program
- Control VR Game on Playground (Placebo Comparator): A relaxing virtual reality game for control group to play in VR playground without training their executive functions
  Interventions: Behavioral: Placebo Virtual Reality Game

INTERVENTIONS:
Behavioral: Virtual Reality-based Interactive Cognitive Training Program — Three virtual reality-based games designed to train inhibitory control, working memory, and cognitive flexibility among children with TBI
  Arms: Virtual Reality games for training executive functions
Behavioral: Placebo Virtual Reality Game — A virtual playground for control group to interact without training executive functions
  Arms: Control VR Game on Playground

SUMMARY:
Childhood traumatic brain injury (TBI) poses significant impairment in children's executive functions (EFs) for moderate to severe injuries, yet interventions specifically designed for children's EF rehabilitation post-TBI and rigorous clinical trials to establish the efficacy of such interventions remain unavailable. In this study, the investigators will conduct a randomized clinical trial to evaluate the efficacy of a novel virtual reality (VR)-based training program for EF rehabilitation for childhood TBI.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a leading cause of acquired disability in U.S. children, with an estimated 700,000 cases every year, presenting in 75% of children with trauma and accounting for 70% of deaths from childhood trauma. Childhood TBIs often result in significant impairment in cognitive functions,1 particularly in core executive functions (EFs) due to the vulnerability of the frontal lobes, especially after a moderate to severe TBI. Core EF is composed of three skills: inhibitory control, working memory, and cognitive flexibility. These skills are associated with impaired EF behaviors, increased attention problems, and lower health-related quality-of-life (HRQOL). However, evidence-based EF rehabilitation programs are lacking. Although a combination of diverse cognitive interventions may improve children's EF, limited affordability, accessibility, adherence, and generalizability hamper clinically adapting and implementing such interventions in the rehabilitation setting. Virtual reality (VR) offers an exciting alternative strategy for EF rehabilitation of childhood TBI due to its flexibility, accessibility, and immersive experiences in three dimensions. These properties may increase adherence to training and foster an enhanced transfer of learned EF skills to untrained tasks in everyday life. Thus far, rigor-ous randomized clinical trials (RCTs) have not been conducted to establish the efficacy of VR-based EF reha-bilitation for childhood TBI.

The overall goal of the project is to assess the efficacy of a novel VR-based interactive cognitive training (VICT) program for EF rehabilitation in children with TBI with the following aims:

Aim 1. Examine VICT's efficacy in improving core and daily EF skills among children with TBI.

Hypothesis 1.1: Children in the intervention group will show enhanced improvement over controls in trained VR-based EF tasks and untrained NIH Toolbox tasks from baseline to post-intervention and follow-up visits; Hypothesis 1.2: The intervention group will show better reported daily EF than controls at the follow-up visit; Hypothesis 1.3: Children in the intervention group will show faster improvement than controls in daily-reported EF skills between post-intervention and follow-up visits.

Aim 2. Examine VICT's efficacy in reducing attentional problems among children with TBI.

Hypothesis 2.1: Children in the intervention group will show a greater reduction in attentional problems as measured by testing on the Conners Continuous Performance Test 3rd Edition™ (Conners CPT 3TM) from baseline to the post-intervention and follow-up visits than controls; Hypothesis 2.2: Children in the intervention group will show fewer everyday attentional problems on the Be-havior Assessment System for Children 3rd Ed (BASC-3) self- and parent-ratings of attention at the follow-up visit than controls; Hypothesis 2.3: The direct effect of the VICT program in reducing attention problems will be mediated by children's EF behaviors as measured by the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2) at the follow-up visit.

Aim 3. Examine VICT's efficacy in improving HRQOL among children with TBI. Hypothesis 3.1: The intervention group will show higher levels of reported HRQOL than controls at follow-up; Hypothesis 3.2: The direct effect of the VICT program on HRQOL at follow-up will be mediated by children's EF skills and ratings of EF behaviors and attention at the post-intervention and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with TBI within the past 12 months and under 18 years at the time of injury;
2. fluent in English; and 3) Score <28 on the Agitated Behavior Scale (if available).

Exclusion Criteria:

1. comorbidities or premorbid disorders that prevent proper administration of VR and study measures,
2. restriction from using electronic devices,
3. post-injury seizure activity.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiabin Shen, PhD, Principal Investigator — University of Massachusetts, Lowell
Locations (2):
- United States (2):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The de-identified datasets and associated documents will be deposited and made available to the public through NICHD Data and Specimen Hub (DASH). DASH has policies and procedures in place that are fully consistent with the NIH Data Sharing Policies and applicable laws and regulations. The final dataset will include demographic and clinical data associated with the nature and severity of patients' injuries, self/parent-reported psychological and behavioral data, performance data on cognitive outcomes. Submitted data will confirm with relevant data and terminology standards as well as policies at NIH, NICHD, and DASH.
Supporting Information: Study Protocol
Time Frame: Data will be deposited to NICHD DASH within one year after the acceptance for publication of the main findings.
Access Criteria: The data will be accessible to the public through NICHD DASH under a carefully-constructed and closely-monitored Data Use Agreement (DUA) following the NICHD DASH DUA template. This will ensure that requesters are (1) committed to using the data shared only for research purposes as approved by the requester's institutional IRB and not to identify any individual participant; (2) committed to securing the data shared using appropriate safety measures and computer technology; (3) committed to not redistribute the shared data to third parties not approved in the DUA, and (4) committed to destroying the data shared after analyses for the intended research are completed, among other measures to ensure the confidentiality of data and protection of subjects' privacy.

REFERENCES:
- [Derived] Shen J, Wang Y, Quinn S, Suskauer SJ, Birch J, Busch T, Svingos A, Crawfis R, Yeates KO, Taylor HG. Efficacy of a virtual reality-based cognitive interactive training program for children with traumatic brain injuries: study protocol for a parallel-group randomized controlled trial. Trials. 2024 Mar 13;25(1):185. doi: 10.1186/s13063-024-08049-1. PMID 38481293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 participants were recruited during 9/2021 and 8/2024 from two participating sites: Spaulding Rehabilitation Hospital and Kennedy Krieger Institute
Period: Overall Study
Arm/Group | Virtual Reality Games for Training Executive Functions | Control VR Game on Playground
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Games for Training Executive Functions | Control VR Game on Playground | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.43 (1.99) | 13.57 (4.20) | 13.00 (3.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 4 | 10
  Black | 1 | 2 | 3
  More than One Race | 0 | 1 | 1
TBI Severity [Count of Participants; unit: Participants] — TBI Severity measured by a categorical variable that classifies a participant as either 'Mild Complicated TBI' or 'Moderate/Severe TBI', as determined by their medical records/physician notes.
  Participants
    Mild Complicated TBI | 3 | 2 | 5
    Moderate/Severe TBI | 4 | 5 | 9
Injury Recency [Mean (Standard Deviation); unit: Days] — Number of Days since Injury
  Days | 73.75 (25.62) | 129.50 (156.64) | 101.62 (108.10)

OUTCOME MEASURES:

1. Primary Outcome: VR-based EF Assessment Task
Description: Performance-based executive function assessment Task in the virtual reality environment built by the research team. There are three tasks within this measurement, each transformed into a z score and summed up to serve as the total score for this measure. A Z-score of 0 in each task represents the sample mean. Higher values represent a better outcome for this measure.
Time Frame: Baseline (at recruitment/before intervention), Post-Intervention (after completion of intervention, up to 2 weeks), Follow-Up (up to 6 months after completion of intervention)
Population: Some participants did not have complete/valid data points for baseline, post, or follow-up visits on this outcome and thus excluded from analysis.
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Virtual Reality Games for Training Executive Functions | Control VR Game on Playground
Number analyzed (Participants) | 6 | 7
Z-Score
  Post Intervention: number analyzed (Participants) | 6 | 6
  Post Intervention | 1.41 (0.77) | 1.53 (0.46)
  Follow Up: number analyzed (Participants) | 5 | 4
  Follow Up | 1.71 (0.59) | 1.82 (0.06)
  Pre Intervention | 1.15 (0.55) | 1.15 (0.34)

2. Secondary Outcome: NIH Toolbox Cognition Battery
Description: Performance-based executive functions tested by three tasks in the NIH Toolbox Cognition Battery: Dimensional Change Card Sort Test, List Sorting Working Memory Test, and Flanker Inhibitory Control and Attention Test. Scores of each task were computed as age-corrected standard scores automatically by the iPad app of the NIH Toolbox Cognition Battery. Each age-corrected standard score is a z-score with a mean of 100 and standard deviation of 15. Total scores are the mean of all three task age-corrected standard scores. Higher scores represent better outcomes.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Virtual Reality Games for Training Executive Functions | Control VR Game on Playground
Number analyzed (Participants) | 6 | 6
Z-score
  Post Intervention: number analyzed (Participants) | 6 | 5
  Post Intervention | 91.11 (11.83) | 90.87 (11.25)
  Follow Up: number analyzed (Participants) | 5 | 4
  Follow Up | 90.87 (11.25) | 88.83 (20.06)
  Pre Intervention | 87.67 (10.26) | 83.56 (12.59)

3. Secondary Outcome: Report-based EF Skills
Description: Behavior Rating Inventory of Executive Function 2; T scores are used (M = 50, SD = 10, no lower/upper limit), T scores from 60 to 64 are considered mildly elevated, and T scores from 65 to 69 are considered potentially clinically elevated. T scores at or above 70 are considered clinically elevated
Time Frame: Follow-Up (up to 6 months after completion of intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Virtual Reality Games for Training Executive Functions | Control VR Game on Playground
Number analyzed (Participants) | 5 | 4
Points
  Parent Report | 52.00 (6.82) | 50.25 (8.81)
  Child Report: number analyzed (Participants) | 4 | 3
  Child Report | 51.75 (12.42) | 49.67 (4.51)

4. Secondary Outcome: Health-related Quality of Life
Description: 23-item PedsQL (Pediatric Quality of Life) Generic Core Scales were designed to measure the core dimensions of health as delineated by the World Health Organization, as well as role (school) functioning. The current study uses its total scores, which is the sum of all 23 items and ranges from 0-100 after transformation. Higher scores indicate better quality of life.
Time Frame: Follow-Up (up to 6 months after completion of intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Games for Training Executive Functions | Control VR Game on Playground
Number analyzed (Participants) | 5 | 4
units on a scale
  Parent Report | 78.88 (20.89) | 75.54 (8.76)
  Child Report | 75.90 (13.49) | 70.67 (4.64)

5. Other Pre Specified Outcome: Motion Sickness
Description: Simulator Sickness Questionnaire, 0-3, higher scores indicate higher levels of motion sickness
Time Frame: Post-Intervention, up to 2 weeks
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Virtual Reality Games for Training Executive Functions | Control VR Game on Playground
Number analyzed (Participants) | 6 | 6
Points | 0.09 (0.13) | 0.24 (0.26)

6. Other Pre Specified Outcome: Perceived Exertion
Description: Borg Perceived Exertion Scale (6-26, higher score indicates greater exertion)
Time Frame: Post-Intervention, up to 2 weeks
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Virtual Reality Games for Training Executive Functions | Control VR Game on Playground
Number analyzed (Participants) | 6 | 6
Points | 7.38 (1.24) | 9.71 (5.06)

7. Other Pre Specified Outcome: Perceived VR Experience
Description: VR User Feedback Survey providing subjective feedback on the VR intervention (1-5, higher scores indicate better VR experience)
Time Frame: Post-Intervention, up to 2 weeks
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Virtual Reality Games for Training Executive Functions | Control VR Game on Playground
Number analyzed (Participants) | 6 | 6
Points
  VR Quality | 2.50 (1.05) | 3.08 (1.28)
  Pleasure | 3.25 (1.33) | 3.92 (1.02)
  motivation-Like to use VR again | 3.17 (0.93) | 3.92 (1.20)
  motivation-use VR in future | 2.83 (1.37) | 3.37 (1.21)
  motivation-use VR in therapies | 3.42 (1.56) | 3.50 (1.52)
  motivation-attend | 3.08 (1.50) | 3.00 (1.67)

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up, up to 6 months after intervention
Description: Any AE or SAE will be reported to the Spaulding Rehabilitation Hospital IRB by site-PI if detected
Arm/Group | Virtual Reality Games for Training Executive Functions | Control VR Game on Playground
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
We encountered significant challenges in patient recruitment during the study period from the pandemic and post-pandemic eras, mostly impacted by significant decrease in available patient volumes as well as shortage and high-turnover of research staff. Recruitment is much lower than anticipated. Therefore, results from this study should be interpreted with caution of the small sample size and variability of the participant characteristics within the sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT04526639/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT04526639/SAP_001.pdf
  • Informed Consent Form (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT04526639/ICF_002.pdf